CLINICAL TRIAL: NCT02073526
Title: Anti-TNF-alpha Trough Level Measurements in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Professor, Oslo University Hospital
Other Study IDs: 2013-1352
Record Dates: First submitted 2014-01-09; First posted 2014-02-27 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Antibodies, Monoclonal; Anti-TNF; TNF-alpha; Trough level; Drug concentration; ELISA
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; Adalimumab; Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anti-TNF: Inflammatory bowel patients age 18 and over treated with anti-TNF agents
  Interventions: Drug: Infliximab, adalimumab, certolizumab pegol

INTERVENTIONS:
Drug: Infliximab, adalimumab, certolizumab pegol — Patients are treated with the above mentioned drugs decided by clinicians

SUMMARY:
Drug serum concentrations will be measured at several time-points for inflammatory disease patients treated with anti-TNF agents. The purpose is to determine which patients that will clinically benefit from either discontinue treatment, adjusting the dose, switch to another anti-TNF agent or a different class of medication.

DETAILED DESCRIPTION:
Crohn´s disease and ulcerative colitis are diseases where the proinflammatory cytokine Tumor Necrosis Factor-alpha (TNF) plays an important role. Anti-TNF agents are used in the treatment. However, some patients do not respond and response rates declines over time. The cause may be immunogenicity against the agent itself, the agent´s failure to neutralize TNF or another biological pathway leading to inflammation. Anti-TNF agents have been administrated as fixed doses at certain frequencies and this may not be optimal for all patients, but recent studies have indicated a correlation between efficacy and serum drug concentration levels (trough levels). Our preliminary data suggest that trough levels early in the treatment course may be predictive of later trough levels. By multiple measurements, this will be assessed. The study will also investigate biological markers in serum and blood cells which may be predictable for trough levels. Finally, we will compare different methods to measure serum drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Inflammatory bowel disease
* Treated with anti-TNF drug
* Follow-up at specialized gastroenterologist in Norway
* Age 18 or over

Exclusion Criteria:

* Patients refusing to participate by not giving their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Inflammatory bowel disease treated with anti-TNF drug
Sampling Method: Non-Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measurement of drug serum concentrations | Serum samples will be collected on average 8 weeks (range 0-90 days) after drug administration
  Drug serum concentration will be measured using an ELISA

SECONDARY OUTCOMES:
Measure soluble TNF-receptor in serum | Measurement will be conducted in 2015 on blood samples stored in a bio-bank
Assay validation | December 2013 - March 2014
  Drug concentration measurements will be conducted with ELISA's with monoclonal and polyclonal antibodies, automated immunofluorometric assay and commercial kits for the purpose to validate tests and establish standards for measurements
Change in individuals drug serum concentration | Serum samples will be collected on average 8 weeks (range 0-90 days) after drug administration
  Intra-individual fluctuations in consecutively measurements during a course of treatment will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Knut EA Lundin, Prof., Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo University Hospital, Oslo, Postboks PB 4950 Nydalen, Norway